CLINICAL TRIAL: NCT07083427
Title: CAPA In-vitro Oocyte Maturation
Brief Title: CAPA In-vitro Oocyte Maturation (CUHK Medical Centre Limited)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CREC-202514
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPA-IVM (Experimental): In CAPA-IVM, the oocyte is treated and matured outside the woman's body, while in classical IVF, the patient is treated. As a consequence, patients undergoing CAPA-IVM are not confronted with the typical risks and burden of systemic ovarian stimulation.
  Interventions: Other: CAPA-IVM

INTERVENTIONS:
Other: CAPA-IVM — In CAPA-IVM, the oocyte is treated and matured outside the woman's body, while in classical IVF, the patient is treated. As a consequence, patients undergoing CAPA-IVM are not confronted with the typical risks and burden of systemic ovarian stimulation.

SUMMARY:
In vitro oocyte maturation (IVM) is a mild-approach assisted reproductive technology (ART). Because of its simplicity, the more favorable financial implications (reduced cost) for patients, and the lower health risk profile of IVM compared to controlled ovarian stimulation (COS) in polycystic ovary syndrome (PCOS) patients, the use of IVM in selected patients may gain increasing interest. Besides its application in patients with polycystic ovaries, IVM technology may have a role in fertility preservation, where young girls and adult women are facing infertility due to gonadotoxic chemotherapeutic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18-50 years old
* Patients seek fertility preservation services
* Patients seek oocyte retrieval services

Exclusion Criteria:

* Patients unable to provide consent/assent (i.e. significant psychiatric problems/cognitive delay)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2035-06-30 (Estimated); Study Completion 2036-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of mature oocytes | 1 week
  Number of mature oocytes after IVM

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided